CLINICAL TRIAL: NCT05413525
Title: Ultrasound-guided Manual Vacuum Aspiration (USG-MVA)
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2021.206
Record Dates: First submitted 2022-05-25; First posted 2022-06-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Ultrasound-guided Manual Vacuum Aspiration; First Trimester Spontaneous Abortion
Keywords: USG-MVA; Ultrasound-guided manual vacuum aspiration; Miscarriage; Cytological analysis; Manual vacuum aspiration
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing USG- MVA for the treatment of early pregnancy loss: Medical notes of all women undergoing USG- MVA for the treatment of early pregnancy loss with gestation < 12 weeks at the Department of Obstetrics and Gynaecology in The Prince of Wales Hospital and Union Hospital will be reviewed.
  Interventions: Procedure: ultrasound-guided manual vacuum aspiration (USG- MVA)

INTERVENTIONS:
Procedure: ultrasound-guided manual vacuum aspiration (USG- MVA) — USG-MVA was carried out as an outpatient day procedure. Women was given a 400μg oral misoprostol tablet 2-3 hours before the procedure. All patients will be given 500mg naproxen orally an hour before the procedure. During the USG-MVA, all the women were placed in the lithotomy position and aseptically dressed. Speculum was performed to visualize the cervix with PCB performed. USG-MVA was performed using a 60ml charged syringe with a flexible curetteattached to it. Transabdominal USG during MVA was performed. During the procedure, local lidocaine gelwas applied to the cervical canal and over the end of the MVA catheter tip during the insertion.The USG-MVA was stopped as soon as USG confirmed that the uterine cavity was empty, defined as a thin endometrial lining with no evidence of retained products of conception.

SUMMARY:
This is a retrospective study to review the current experience of USG-MVA in Hong Kong and also evaluate the effectiveness of USG-MVA in cytological analysis in the management of first trimester miscarriage.

DETAILED DESCRIPTION:
Miscarriage can be managed expectantly, medically or surgically. In cases where cytogenetic analysis is wanted, surgical evacuation is the ideal option as the POC is difficult to be obtained after medical evacuation. However, traditional surgical evacuation requires the procedure to be performed under general anesthesia using an electric vacuum aspiration (EVA). Moreover, the chorionic villi obtained via POC is often less intact and dispersed, making the identification and analysis difficult. Manual vacuum aspiration (MVA) was first introduced in 1973. The procedure is performed using a hand-held 60ml syringe to create the suction force and the intrauterine contents are aspirated using either a flexible or rigid cannula attached on it. The procedure can be performed in an outpatient setting with simple oral analgesics or conscious sedation given beforehand.

The investigators have previously evaluated the acceptability and feasibility of the addition of ultrasound guidance during the procedure. The investigators found that ultrasound-guided manual vacuum aspiration (USG-MVA) is an effective alternative treatment modality to medical and traditional surgical evacuation under general anesthesia for the management of first trimester delayed or incomplete miscarriage. The procedure has been introduced in our locality since 2015. Since then, the investigators have performed more than 200 cases of USG-MVA locally. However, the subsequent local experience of USG-MVA and culture failure rate in the POC during cytological analysis obtained via this method remains limited in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or above
* Women with miscarriage who are suitable candidates for USG-MVA
* first trimester delayed miscarriage ≤ 12 weeks of gestation
* incomplete miscarriage with POG ≤ 5cm
* hemodynamically stable
* tolerates well with speculum examination

Exclusion Criteria:

* Women who are not feasible for the USG-MVA
* cervical stenosis
* fibroid uterus ≥12 weeks in size
* known uterine malformation
* bleeding disorder
* suspicion of active infection
* inability to tolerate pelvic examination
* History of allergy to misprostol or same group of medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with first trimester miscarriage
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
complete evacuation rate of the products of conception | Three weeks from surgery to follow-up
  To evaluate the effectiveness in terms of the complete evacuation rate of the products of conception in patients undergoing USG-MVA in the treatment of first trimester miscarriage

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Three weeks from surgery to follow-up
  To assess the complications in patients undergoing the USG-MVA procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Chinese University of Hong Kong, Hong Kong, Shatin
  - Union Hospital, Hong Kong